CLINICAL TRIAL: NCT00247468
Title: Strict Glucose Control of Pediatric ICU Patients to Reduce Mortality and Morbidity
Brief Title: Strict Glucose Control of Pediatric Intensive Care Unit (ICU) Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never received IRB approval
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-2-3160
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Respiratory Failure; Cardiovascular Failure; Sepsis; Trauma
MeSH Terms: conditions — Respiratory Insufficiency; Sepsis; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Strict Glucose Control

SUMMARY:
The study objective is to improve morbidity and mortality of high-risk critically ill children. Our hypothesis is that a strict ICU glucose control protocol will decrease morbidity and mortality associated with hyperglycemia in a population of high-risk critically ill pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Vasoactive infusion (e.g. dopamine, epinephrine, norepinephrine) and/or
* Invasive mechanical ventilation
* Age between 1 mo and 21 yrs

Exclusion Criteria:

* Type I diabetes mellitus
* Have an illness that requires insulin daily
* Recipients of solid organ transplants
* Participation in an experimental trial that might affect outcome
* Post-operative patients with planned extubation upon recovery
* Patients on a dopamine infusion of less than 3 mcg/kg/minute

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2004-12 (Actual); Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
30-day mortality rate from the time of enrollment

SECONDARY OUTCOMES:
Pediatric Overall Performance Category scores at ICU discharge and 6 months post-discharge
rates of nosocomial bloodstream infections
time to resolution of organ failure (mechanical ventilator days and days of vasopressor support)
change in Pediatric Logistic Organ Dysfunction scores
requirement of dialysis or hemofiltration for patients with acute renal failure
volume of blood product transfusions per kilogram body weight (vol/kg).

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Nadkarni, MD, Principal Investigator — Children's Hospital of Philadelphia

IPD SHARING:
Plan to Share IPD: No